CLINICAL TRIAL: NCT01022515
Title: Clinical Application of New Pheochromocytoma Markers: INSERM Pilot Study of the Specificity of Elevated Plasma EM66 Concentrations in Patients With Pheochromocytoma or Paraganglioma Compared to Patients With Essential Hypertension
Brief Title: Specificity of Elevated Plasma EM66 Levels in Pheochromocytoma
Acronym: PHEO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Rouen (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2007/081/HP; 2007-AO1004-49 (Registry Identifier: RCB)
Record Dates: First submitted 2009-11-17; First posted 2009-12-01 (Estimated); Last update posted 2026-02-06 (Actual); Status verified 2014-06

CONDITIONS: Pheochromocytoma; Paraganglioma; Essential Hypertension
Keywords: pheochromocytoma; paraganglioma; hypertension
MeSH Terms: conditions — Pheochromocytoma; Paraganglioma; Essential Hypertension; Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- patients with pheochromocytoma (Other): Patients with pheochromocytoma / paraganglioma are being followed as recommended according to international standards. No intervention is expected except regular measurement of plasma CgA (as usual) and EM66 (research purpose) levels.
  Interventions: Other: usual follow up with regular EM66 & Cga levels assessment
- Patients with essential hypertension (Other): Patients with essential hypertension will be selected as controls. EM66 and CgA plasma levels will be assessed in these patients after having excluded the presence of a pheochromocytoma / paraganglioma with normal urinary metanephrines / normetanephrines excretion levels.
  Interventions: Other: plasma EM66 & CgA levels assessment

INTERVENTIONS:
Other: plasma EM66 & CgA levels assessment — After inclusion checking to eliminate the presence of pheochromocytoma / paraganglioma, a blood sample will be drawn to assess plasma EM66 and CgA levels.
  Arms: Patients with essential hypertension
Other: usual follow up with regular EM66 & Cga levels assessment — Patients with pheochromocytoma / paraganglioma will be followed-up as the international standards recommend.
  Regularly, blood samples will be drawn for the usual assessment of CgA levels and also EM66 (research purpose) levels.
  Arms: patients with pheochromocytoma

SUMMARY:
Pheochromocytoma or paraganglioma are tumors generating hypertension as a symptom. Different biological tests are currently available to diagnose these tumors. However, they all lack specificity since they do not distinguish cases of hypertension without pheochromocytoma or paraganglioma. To improve the diagnostic specificity of these tumors, the investigators are testing a new marker called EM66.

DETAILED DESCRIPTION:
Neuroendocrine tumors (NT) correspond to neoplasms that develop from endocrine and neuroendocrine cells scattered throughout the body. They are characterized by the occurrence, in their cytoplasm, of dense-core secretory vesicles containing hormones, neuropeptides and acidic proteins such as granins. The diversity of NT (from hypophysis, pancreas, adrenal, gastrointestinal tract) makes very difficult the identification and evaluation of the different types of tumors by the diagnostic and prognostic tools currently available. We have thus established a research program aimed at identifying new biological markers for the detection, the prognosis and the follow-up of NT by seeking in tumor and plasma samples of patients, granin-derived peptides. Our program was initiated on one type of NT : pheochromocytoma. These neoplasms correspond to tumoral chromaffin cells mainly originating from the adrenal medulla. It is considered that 10 % of pheochromocytoma patients will develop metastases and, currently, except in the presence of metastases, there are no means to predict malignancy of the tumor. We setup a radioimmunoassay of EM66 (a secretogranin II-derived peptide) that allowed us to demonstrate that (i) plasma concentrations of the peptide are significantly elevated in pheochromocytoma patients, (ii) combined with other biological tests EM66 measurement increase the diagnostic sensitivity for these neoplasms, (iii) after surgical removal of the tumor, plasma EM66 concentrations rapidly return to basal level and, (iv) intra-tumoral EM66 concentrations are higher in benign than in malignant pheochromocytomas (Yon et al., 2003, Guillemot et al., 2006). These results reveal that EM66 constitutes a novel tool for the diagnosis, prognosis and follow-up of pheochromocytoma. In the frame of a clinical use of an EM66 measurement test, it is necessary to evaluate the specificity of this marker. For instance, renal deficiency, hypergastrinemia, reduction of renal clearance, type A gastritis, Crohns disease, or proton-pump inhibitory treatment, lead to increase plasma chromogranin A (CgA) concentrations (false-positive cases). In addition, while hypertension account for one of the symptoms of pheochromocytoma patients, in essential hypertensive patients, CgA levels are higher than in normotensive individuals. The main objective of our clinical transfer research project consists to study the specificity of the measurement of EM66 as a diagnostic and prognostic marker of pheochromocytoma. This multicentric study will allow us to compare plasma EM66 levels in pheochromocytoma patients with a cohort of essential hypertensive patients. At the same time, in a long-range prospect, due to the lack of malignancy markers for these tumors, we will investigate if plasma or tumor EM66 levels are correlated to the differentiation status of pheochromocytomas, and if the expression level of a set of genes that we identified by a transcriptomic approach developed in the laboratory, is associated with the malignant status of the tumors. The stakes of this transfer research, involving our laboratory and the Center for Clinical Investigations (CIC) of Rouen and Lille, are to provide an easy and simple novel tool to practitioners and anatomo-pathologists for the screening, the evaluation and the follow-up of patients with neuroendocrine tumors.

ELIGIBILITY:
Patients with pheochromocytoma/paraganglioma

Inclusion criteria :

* men & women, age > 18 years old
* Newly diagnosed patient : suspicion of pheochromocytoma or paraganglioma with elevation of urinary metanephrines and/or normetanephrines along with evidence of tumor which surgical removal is considered (histological findings following surgery will be the gold standard for final diagnosis and inclusion in the study)
* During follow-up of a patient with known genetic predisposition to pheochromocytoma/paraganglioma : suspicion of pheochromocytoma or paraganglioma with or without elevation of urinary metanephrines and/or normetanephrines along with evidence of a tumor which surgical removal is considered (histological findings following surgery will be the gold standard for final diagnosis and inclusion in the study) ,
* Patients with known pheochromocytoma/paraganglioma, whether malignant or not, whether with metanephrine secretion or not, With tumor sites at inclusion in the study
* Patients informed and willing to participate in the study
* Patients with medical insurance (French social security) Non inclusion criteria
* Patients newly diagnosed, recently operated and the histological findings disprove pheochromocytoma or paraganglioma.
* patient imprisoned or under legal protection.

Patients with essential hypertension Inclusion criteria

* men & women, age > 18 years old
* paired with a patient with pheochromocytoma/paraganglioma for : gender, age (± 5 years) and centre
* patient with hypertension. No aetiology was found after initial check up.
* Normal 24 hours urinary excretion of metanephrines & normetanephrines
* For women of childbearing potential : effective contraceptive method and negative urinary pregnancy test
* Patients informed and willing to participate in the study
* Patients with medical insurance (French social security) Non inclusion criteria
* Treatment with proton-pump inhibitors in the 8 days before inclusion in the study
* Treatment with beta-blockers, antidepressants, Benzodiazepins, dopa, alphamethyl dopa, if this treatment cannot be interrupted during the study (i.e. for approximately 10 days)
* patient imprisoned or under legal protection.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2008-11; Primary Completion 2022-04-13 (Actual); Study Completion 2022-04-13 (Actual)

PRIMARY OUTCOMES:
Plasma EM66 | two years

SECONDARY OUTCOMES:
Plasma Chromogranin A levels | before treatement

CONTACTS AND LOCATIONS:
Overall Officials: Anne F Cailleux, MD, Principal Investigator — University Hospital, Rouen
Locations (8):
- France (8):
  - CIC 9301, Lille
  - Endocrinology Department, Lille
  - Inserm U982/EA 4310; Rouen University (DC2N), Mont-Saint-Aignan
  - Cardiology Department, Paris
  - CIC 9304, Paris
  - Cic-Crb 0204, Rouen
  - Endocrinology Department, Rouen
  - Endocrinology Department, Gustave-Roussy Institute, Villejuif